CLINICAL TRIAL: NCT00872183
Title: Exploring a Motor Learning Technique Based on the Mirror Motor Neuron System
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 090098; 09-N-0098
Record Dates: First submitted 2009-03-28; First posted 2009-03-31 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2012-05-03

CONDITIONS: Healthy
Keywords: Motor Learning; Mirror Neurons; Healthy Volunteer; HV

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Background:

* Techniques that teach finger movements are commonly used to explore how humans learn to move. Researchers have designed a simple, new method of learning finger movements, which will be explored for the first time in this study. The method is based on how individuals mimic other people's movements.
* Previous studies have shown that a brain protein called brain-derived neurotrophic factor (BDNF) may be important in movement and in learning. There are normal variations in the gene for BDNF. As an optional component, this study will also look at whether these gene variations are associated with differences in movement learning.

Objectives:

* To compare the new motor learning technique with a classic technique to test its usefulness.
* To examine whether genetic variations have an effect on motor learning.

Eligibility:

* Healthy volunteers between the ages of 18 and 50, who are right-handed.

Design:

* The study will involve two visits to the National Institutes of Health Clinical Center.
* Visit 1: Medical and neurologic examination to determine whether the volunteer is eligible to participate further in the study. This screening visit will take about 1 hour.
* Visit 2: Volunteers will perform a motor learning task by interacting with a computer program. In response to images on the computer monitor, volunteers will press buttons on the keyboard as quickly and accurately as possible. The motor learning task will last up to 3 hours.
* If a volunteer agrees to genetic testing, researchers will also draw blood for study. Genetic testing is not required to participate in the motor learning parts of the study.

DETAILED DESCRIPTION:
Objective

Humans develop skilled movements such as using a spoon or dancing a waltz through a process known as "motor learning. Harnessing this innate process for its therapeutic potential is an attractive strategy to help patients suffering from diseases of movement disorders, yet we do not yet fully understand the normal phenomenon. This study will utilize new paradigms to explore the physiology of motor learning. It will test the validity of a traditional motor learning task that has been modified to invoke the mirror neuron system and odor conditioning. Additionally, by taking advantage of the unique opportunity to assess motor learning awareness immediately following the task, it will also explore this behavioral-cognitive relationship. Thus, this work will lay the foundation for further physiologic characterization of a novel motor learning technique and may support the development of future therapies.

Study Population

We will study up to one hundred fifty-two healthy, right-handed volunteers who are 18 to 50 years old.

Design

In phase I of the study, volunteers will be seated in front of a computer monitor with their right hands on a keyboard and respond to visual cues presented on the monitor by pressing the associated, finger-specific keys as quickly and accurately as possible. Each volunteer will be presented only the standard visuospatial or the novel mirror cues, defining the two reaction time task paradigms and experimental groups. In phases II and III of the study, a similar task will take place while subjects undergo magnetic resonance imaging scanning either in the presence or absence of an odor. In addition to the motor learning tasks above, volunteers will have the option to participate in genetic testing for normal genetic variability that may affect motor learning.

Outcome Measure

The primary outcomes are motor learning and awareness, which will be measured by the key-press reaction time and accuracy, respectively.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Age 18-50 years
* Right-handedness

EXCLUSION CRITERIA:

* Arthritis or other physically limiting disability, amputation, or significant trauma of either hand
* Professional musician or stenographer
* Persistent neurologic deficit of cognition, movement, or sensation or any history of a central nervous system lesion
* Regular use of any neurotropic or psychotropic medication (e.g., narcotic analgesic, anxiolytic, anti-histamine) or any use within twenty-four hours of the motor learning task.
* Blindness or visual acuity lower than necessary to distinguish visual stimuli on the display monitor
* Impaired decisional capacity or inability to provide informed consent
* Previous experience with a serial reaction time task type of study
* Nasopharyngeal illness, injury, or dysfunction (Phase III only)
* Inability to smell odorized air during screening exam (Phase III only)
* Pregnancy (Phases II and III only)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 76 (Actual)
Dates: Start 2009-03-25; Study Completion 2012-05-03

CONTACTS AND LOCATIONS:
Overall Officials: Bibiana Bielekova, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Abrahamse EL, Verwey WB. Context dependent learning in the serial RT task. Psychol Res. 2008 Jul;72(4):397-404. doi: 10.1007/s00426-007-0123-5. Epub 2007 Aug 3. PMID 17674034
- [Background] Ashe J, Lungu OV, Basford AT, Lu X. Cortical control of motor sequences. Curr Opin Neurobiol. 2006 Apr;16(2):213-21. doi: 10.1016/j.conb.2006.03.008. Epub 2006 Mar 24. PMID 16563734
- [Background] Bird G, Osman M, Saggerson A, Heyes C. Sequence learning by action, observation and action observation. Br J Psychol. 2005 Aug;96(Pt 3):371-88. doi: 10.1348/000712605X47440. PMID 16131413